CLINICAL TRIAL: NCT03679117
Title: Prenatal Mindfulness Training for Pregnant Women at Risk for Hypertension
Brief Title: Prenatal Mindfulness & Hypertension Study
Acronym: HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Margaret Bublitz, Research Scientist, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1303286; P20GM103652 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-09-20 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Hypertension in Pregnancy
Keywords: mindfulness; pregnancy; hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized trial in which participants are assigned to mindfulness training or treatment as usual.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental): Phone-delivered mindfulness training
  Interventions: Behavioral: Mindfulness Training
- Treatment as Usual (No Intervention): Prenatal care

INTERVENTIONS:
Behavioral: Mindfulness Training — Phone-delivered mindfulness training. 8 weeks of 30 minute phone sessions with an instructor, plus 15 minutes of self-guided practice.
  Arms: Mindfulness Training

SUMMARY:
Hypertensive disorders of pregnancy are one of the greatest causes of death to mothers and babies. These disorders affect 1 out of every 10 pregnancies, the rate is increasing in the United States, and rate of recurrence is as high as 50%. Treatments to prevent hypertensive disorders of pregnancy from happening in future pregnancies are limited. There are currently no effective interventions to prevent hypertension recurrence in pregnancy that do not involve medications.

Mindfulness interventions hold great potential as a medication-free approach to prevent the recurrence of hypertension in pregnant women with histories of hypertensive disorders. However, traditional group-based mindfulness training interventions, requiring 2.5 hours of class attendance for 8 weeks plus a full-day retreat, are very difficult for pregnant women with medical conditions to attend.

The goal of the current study is to determine if phone-delivered mindfulness training is an acceptable intervention among pregnant women with histories of hypertensive disorders of pregnancy. 20 pregnant women with histories of hypertensive disorders of pregnancy will be randomly picked to participate in an 8-week phone-delivered mindfulness training intervention (N=10) or usual care (N=10). All women will undergo blood pressure monitoring before and after the intervention. The investigators predict that phone-delivered mindfulness training will reduce risk for hypertension recurrence.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy are one of the greatest causes of perinatal morbidity and mortality. Hypertensive disorders of pregnancy affect 1 out of every 10 pregnancies, the rate has increased substantially over the past several decades, and rates of recurrence are as high as 50%. Treatments to prevent the recurrence of hypertension are extremely limited and include watchful waiting, anti-hypertensive medications, or ultimately, early delivery. There are currently no effective alternatives to pharmacological interventions to prevent hypertension recurrence in pregnancy.

Mindfulness interventions hold great potential as a non-pharmacological approach to reduce stress and prevent the recurrence of hypertension in pregnant women with histories of hypertensive disorders. However, traditional group-based mindfulness training interventions, requiring 2.5 hours of class attendance for 8 weeks plus a full-day retreat, are infeasible in pregnancies complicated by hypertensive disorders due to the need for activity restriction, hospitalization, and increased maternal and fetal monitoring.

The goal of the current study is to determine if phone-delivered mindfulness training is feasible and acceptable among pregnant women with histories of hypertensive disorders of pregnancy. 20 pregnant women with histories of hypertensive disorders of pregnancy will be randomized to an 8-week phone-delivered mindfulness training intervention (N=10) or usual care (N=10). All women will undergo 24-hour ambulatory blood pressure monitoring before and after the intervention. The investigators will used a mixed-methods approach using both quantitative and qualitative data to examine feasibility/acceptability. The working hypothesis, to be tested in a fully-powered randomized controlled trial, is that phone-delivered mindfulness training will reduce risk for hypertension recurrence.

ELIGIBILITY:
Inclusion criteria:

* > 18 years old,
* Singleton pregnancy,
* English speaking,
* <20 weeks' gestation at enrollment,
* History of a hypertensive disorder in a prior pregnancy.

Exclusion criteria:

* No current engagement in mindfulness training (defined as weekly yoga, mindfulness exercises (including on-line), or meditation).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Bublitz, PhD, Principal Investigator — Women's Medicine Collaborative
Locations (1):
- Women's Medicine Collaborative, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bublitz MH, Anderson M, Bourjeily G, Salmoirago-Blotcher E. Psychological mechanisms of prenatal mindfulness training on antenatal blood pressure reduction: A pilot study. J Psychosom Res. 2025 Aug;195:112183. doi: 10.1016/j.jpsychores.2025.112183. Epub 2025 Jun 6. PMID 40505593
- [Derived] Sharp M, Ward LG, Pomerantz M, Bourjeily G, Guthrie KM, Salmoirago-Blotcher E, Desmarattes A, Bublitz MH. Prenatal Mindfulness Training and Interoceptive Awareness in Pregnant People at Risk for Hypertensive Disorders. J Integr Complement Med. 2024 Dec;30(12):1200-1208. doi: 10.1089/jicm.2024.0121. Epub 2024 Jul 8. PMID 38976481
- [Derived] Unger KG, Sanapo L, Bourjeily G, Salmoirago-Blotcher E, Bublitz MH. The Impact of Mindfulness Treatment on Maternal Inflammation and Fetal Neurodevelopment Among Participants with Histories of Hypertensive Disorders. J Integr Complement Med. 2024 Jan;30(1):85-89. doi: 10.1089/jicm.2023.0254. Epub 2023 Sep 26. PMID 37751286
- [Derived] Bublitz MH, Salmoirago-Blotcher E, Sanapo L, Ayala N, Mehta N, Bourjeily G. Feasibility, acceptability, and preliminary effects of mindfulness training on antenatal blood pressure. J Psychosom Res. 2023 Feb;165:111146. doi: 10.1016/j.jpsychores.2023.111146. Epub 2023 Jan 5. PMID 36621212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew prior to randomization. This is why 30 participants were enrolled and 29 randomized.
Groups:
- Treatment as Usual: Usual prenatal care to prevent and treat hypertension
Period: Overall Study
Arm/Group | Mindfulness Training | Treatment as Usual
Started | 15 | 14
Completed | 12 | 14
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training | Treatment as Usual | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4) | 32 (5) | 32 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 11 | 9 | 20
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 117 (11) | 125 (14) | 121 (13)

OUTCOME MEASURES:

1. Primary Outcome: Retention and Adherence
Description: Number of participants that completed greater than 5 mindfulness sessions or completed the follow up interview.
Time Frame: Through study completion, an average of 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training | Treatment as Usual
Number analyzed (Participants) | 15 | 14
Participants | 12 | 11

2. Secondary Outcome: Hypertension Diagnosis
Description: Number of participants with a diagnosis of hypertensive disorders of pregnancy
Time Frame: Through study completion, an average of 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training | Treatment as Usual
Number analyzed (Participants) | 15 | 14
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during participation in the RCT approximately 20 weeks.
Arm/Group | Mindfulness Training | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 8/15 | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training (N=15) | Treatment as Usual (N=14)
Suicidal ideation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
High blood pressure (Blood and lymphatic system disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03679117/Prot_SAP_ICF_001.pdf